CLINICAL TRIAL: NCT02261194
Title: Effect of a Self-care Intervention on Depression in People With Age-related Macular Degeneration or Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); Fondation Antoine Turmel (Unknown)
Responsible Party: Principal Investigator, Ellen Freeman, Associate Professor, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Réseau Vision Freeman
Record Dates: First submitted 2014-10-02; First posted 2014-10-10 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Depression; Age-related Macular Degeneration
Keywords: depression; age-related macular degeneration; self-care; self-help
MeSH Terms: conditions — Depression; Macular Degeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Care Tools (Experimental): The tool binder includes 3 core tools and 4 supplemental tools. The tools that will be provided include a variety of self-care approaches to manage depression including audio-visual, internet, and paper-based tools that might appeal to individuals with different learning styles. The 3 core tools consist of the Antidepressant Skills Workbook, a Mood Monitoring Tool, and a DVD on depression.
  Interventions: Behavioral: Self-Care Tools
- Delayed Self-Care Tools (No Intervention): This group will receive the self-care tools at the conclusion of the study.

INTERVENTIONS:
Behavioral: Self-Care Tools
  Arms: Self-Care Tools

SUMMARY:
The purpose of this trial is to determine the short-term effect of a self-care intervention on depression in patients with age-related macular degeneration or diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of wet or dry AMD or diabetic retinopathy
* age 50 years and older
* at least mild depressive symptoms (a score of 5 or more on the PHQ-9)
* no legal blindness (visual acuity better than 20/200 in better eye).

Exclusion Criteria:

* the current use of cognitive behavioural therapy
* suicidal intent
* ocular surgery during the study period (intravitreal anti-VEGF injections will be allowed, e.g. Lucentis)
* cognitive impairment
* inability to speak and understand French or English
* profound hearing impairment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms | Baseline and 8 weeks
  Depressive symptoms will be measured by the PHQ-9, a validated 9 item instrument.

SECONDARY OUTCOMES:
Change in severity of anxiety symptoms | Baseline and 8 weeks
  The GAD-7 can be used to establish probable diagnoses of generalized anxiety disorder as well as grade its severity (mild, moderate and severe).
Change in self-efficacy | Baseline and 8 weeks
  Self-efficacy will be measured with a 4-item scale, adapted from a validated diabetes self-care self-efficacy scale. Scores range from 0-12.
Change in life space | Baseline and 8 weeks
  The Life Space Assessment asks about the spatial extent in which the participant has traveled over the last month. Scores range from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E. Freeman, PhD, Principal Investigator — Maisonneuve-Rosemont Hospital and University of Montreal
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada